CLINICAL TRIAL: NCT05362253
Title: The Effect of Micro-Conjunctival Autografting Combined With Amniotic Membrane Transplantation on Treating Recurrent Pterygium: A Non-randomized Controlled Trial
Brief Title: Micro-Conjunctival Autografting Combined With Amniotic Membrane Transplantation Treating Recurrent Pterygium Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yifeng Yu (Other)
Responsible Party: Sponsor-Investigator, Yifeng Yu, Associate professor, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2021]NO.(024)
Record Dates: First submitted 2022-04-26; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Recurrent Pterygium; Micro-Conjunctival Autografting Combined With Amniotic Membrane Transplantation
Keywords: Recurrent pterygium; Conjunctival flap; Transplantation
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group received micro-conjunctival autograft combined with amniotic membrane transplantation.
  Interventions: Procedure: Micro-Conjunctival Autograft Combined with Amniotic Membrane Transplantation
- control group (Active Comparator): The control group received given routine autologous conjunctival transplantation.
  Interventions: Procedure: Conventional Autologous Conjunctival Transplantation

INTERVENTIONS:
Procedure: Micro-Conjunctival Autograft Combined with Amniotic Membrane Transplantation — 1. Disinfection, anaesthesia and excision of recurrent pterygium are the same as conventional autologous conjunctival transplantation.
  2. The biological freeze-dried amniotic membrane (Jiangxi Ruiji Biological engineering technology Co., Ltd., Nanchang, China), equivalent in size to the exposed scleral surface, was flat mounted on the exposed scleral area , and the amniotic membrane was fixed on the superficial sclera with 10-0 suture.
  3. After amniotic membrane graft was fixed, 2% lidocaine was applied to the superior temporal conjunctiva.
  4. Take the conjunctival epithelial graft with the length equivalent to the neck of recurrent pterygium and the width of 1.5mm ~ 2.0mm, and translate it on amniotic membrane surface near corneal limbus. The conjunctival flap was secured with 10-0 suture.
  5. Last, tobramycin and dexamethasone eye ointment was applied and bandaged with dressing.
  Arms: experimental group
Procedure: Conventional Autologous Conjunctival Transplantation — 1. Routine disinfection and anaesthesia.
  2. To bluntly separate and excise pterygium.
  3. Remove pterygium tissue on the corneal surface with a round blade.
  4. Place a cotton ball slightly infiltrated with diluent Bleomycin A5 Hydrochloride for Injection on the exposed sclera for 1 minute and flushed away later.
  5. After anesthesia, take the superior temporal conjunctival epithelium equal to the size of the exposed scleral and translate it to the exposed scleral surface (the limbus side of the graft corresponds to the limbus of the graft bed), and fixed with 10-0 suture.
  6. The free conjunctival margin of the conjunctival flap sampling area was sutured intermittently with 10-0 suture.
  7. Apply tobramycin dexamethasone eye ointment and wrap the eyes with dressing after operation.
  Arms: control group

SUMMARY:
To observe the effect of micro-conjunctival autografting combined with amniotic membrane transplantation on the postoperative recurrence, complications and ocular surface symptoms among patients with recurrent pterygium.

DETAILED DESCRIPTION:
Recurrent pterygium is a common postoperative complication of pterygium surgery, the postoperative recurrence rate is about 1.44% and needs careful treatment. At present, surgical is the main and most effective treatment of recurrent pterygium. Among various surgical methods, autologous conjunctival transplantation is regarded as the first choice in normal conditions. However, the scope of conjunctival transplantation is positively correlated with the degree of ocular surface damage. Therefore, our research aimed to use micro conjunctival transplantation（1.5mm×3.0mm） to reconstruct limbal conjunctiva and amniotic membrane to cover the whole pterygium resection area to better protect conjunctival sac and ocular surface.

ELIGIBILITY:
Inclusion Criteria:

1. age⩾18;
2. relapsed after pterygium surgery once;
3. invading the cornea 2.00~5.00mm.

Exclusion Criteria:

1. having obvious severe systemic organic diseases and mental diseases;
2. In lactation or pregnancy or planned pregnancy;
3. combined with eye diseases such as severe eyelid insufficiency, dry eye, chemical injury of cornea and conjunctiva, etc.;
4. used drugs that may affect the growth and metabolism of corneal epithelium within four weeks before inclusion in the study;
5. received pterygium surgery twice or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Changes of grade of conjunctival hyperplasia | Day 0#3#7 and14, Month 1#3 and 6.
  Grade 1, no significant difference from normal eyes (no recurrence); Grade 2, a little episcleral vessels in the pterygium excision area, which extends to the corneoscleral limbus but does not exceed, and there is no fibrous tissue hyperplasia (no recurrence); Grade 3, having proliferative fibrous tissue in the resection area, which does not exceed the limbus (no recurrence); Grade 4, the cornea is invaded by proliferative fibrous tissue, and this grade is true pterygium recurrence (recurrence).
Changes of Schirmer test I | Day 0#3#7 and14, Month 1#3 and 6.
  5-minute Schirmer test I
Changes of ocular surface symptom scores | Day 0#3#7 and14, Month 1#3 and 6.
  Include dryness, burning, foreign body and pain sensation. The full score of each symptom is 100 points, with a score of 0 reflecting no discomfort, 100 was considered as the maximum discomfort.

SECONDARY OUTCOMES:
Changes of corneal epithelial repair time | Day 0#3#7 and14, Month 1#3 and 6.
  Corneal fluorescein sodium staining was applied to assess the epithelial repair after operation.
Changes of visual acuity | Day 0#3#7 and14, Month 1#3 and 6.
  To observe the changes of visual acuity around operation.

OTHER OUTCOMES:
Changes of pterygium size | Day 0#3#7 and14, Month 1#3 and 6.
  The pterygium size is recorded by the longest length of its invasion into the cornea.
Changes of intraocular pressure | Day 0#3#7 and14, Month 1#3 and 6.
  To monitor intraocular pressure during the period of useing glucocorticoids.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No